CLINICAL TRIAL: NCT04258046
Title: Phase II Clinical Trial of MEK Inhibitor Trametinib in the Treatment of Complicated Extracranial Arterial Venous Malformation (VM)
Brief Title: Trametinib in the Treatment of Complicated Extracranial Arterial Venous Malformation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Joyce Teng, Director of Pediatric Dermatology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53105
Record Dates: First submitted 2020-01-16; First posted 2020-02-06 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Venous Malformation; Arterial Disease
MeSH Terms: interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Trametinib (Experimental): Patients will receive oral trametinib once daily
  Interventions: Drug: Trametinib tablet

INTERVENTIONS:
Drug: Trametinib tablet — Drug is supplied in 0.5 mg and 2 mg tablets

SUMMARY:
Arteriovenous malformation (AVM) is a congenital vascular anomaly that progresses throughout life and causes complications including tissue destruction due to rapid overgrowth, bleeding, functional deficits, severe deformity and cardiac failure. Unfortunately, traditional managements have transient benefits with more than 90 recurrence rate within a year. Therefore, there is a significant unmet medical need. The purpose of this study is to assess the safety and efficacy of Trametinib in children and adults with Extracranial Arteriovenous Malformation (AVM).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 12 years and ≤ 60 years
* Confirmed diagnosis of complicated extracranial AVMs made by a physician who is familiar with this condition.
* Genetic testing for mutations within MAP2K1 or remaining RAS/MAPK pathway is preferred but not mandatory
* Patient is able to swallow and/or retain oral medication via G tube
* All clinical and laboratory studies to determine eligibility will be performed within six weeks prior to enrollment unless otherwise indicated.
* Patients who have undergone surgical resection or interventional radiology procedures (sclerotherapy) of their AVM are eligible if they meet all inclusion criteria after these procedures
* At least 4 weeks from undergoing any major surgery
* Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* Myelosuppressive chemotherapy: None within 4 weeks of entry into this study.
* At least 14 days since the completion of therapy with a biologic. For agents that have known adverse events occurring beyond 14 days after administration, this period must be extended beyond the time during which adverse events are known to occur. These patients must be discussed among PI and other investigators on a case-by-case basis.
* Patients must not have received an investigational drug within the prior 4 weeks.
* Not within 6 months prior to entering study if AVM is within field of radiation

Exclusion Criteria:

* AVM due to germline mutation such as PTEN
* Prior MEK inhibitor therapy or have allergy or contraindication to MEK inhibitor
* Unable to swallow PO drugs or administer the drug via G tube
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study treatment or who have not recovered from side effects of such procedure
* Patients with evidence of or history of cardiovascular risk
* Patients with retinal vein occlusion, hemorrhage or have a history of such conditions.
* Patients who are currently on other immunosuppressive medication(s)
* Patients who have an uncontrolled infection
* Unstable health status that may interfere with completing study
* Unable to travel to clinic as requested
* Patients unwilling or unable to comply with the protocol, or who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Females of child-bearing potential must be willing to practice acceptable methods of birth control.
* Additionally, females of childbearing potential must have a negative serum pregnancy test result from 7 days prior to the initiation of the medication to 3 months after the final administration of the medication. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the period when they are receiving the study drug and for 3 months thereafter.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease response rate by investigator assessment at Month 6 | Month 6
  Combining a composite of radiographic, clinical, functional impairment, and quality of life measures.

SECONDARY OUTCOMES:
Change from baseline in MRI Volumetric Scan Measurement of Targeted Disease Area | Month 6
Change from baseline in MRI Volumetric Scan Measurement of Targeted Disease Area | Month 12
Disease response rate by investigator assessment at Month 12 | Month 12
  Combining a composite of radiographic, clinical, functional impairment, and quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Teng, MD, PhD, FAAD, Principal Investigator — Stanford University
Locations (1):
- Pediatric Dermatology Clinic at Stanford Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu AS, Mulliken JB, Zurakowski D, Fishman SJ, Greene AK. Extracranial arteriovenous malformations: natural progression and recurrence after treatment. Plast Reconstr Surg. 2010 Apr;125(4):1185-1194. doi: 10.1097/PRS.0b013e3181d18070. PMID 20335868
- [Background] Couto JA, Huang AY, Konczyk DJ, Goss JA, Fishman SJ, Mulliken JB, Warman ML, Greene AK. Somatic MAP2K1 Mutations Are Associated with Extracranial Arteriovenous Malformation. Am J Hum Genet. 2017 Mar 2;100(3):546-554. doi: 10.1016/j.ajhg.2017.01.018. Epub 2017 Feb 9. PMID 28190454
- [Background] Goss JA, Konczyk DJ, Smits PJ, Kozakewich HPW, Alomari AI, Al-Ibraheemi A, Taghinia AH, Dickie BH, Adams DM, Fishman SJ, Mulliken JB, Warman ML, Greene AK. Intramuscular fast-flow vascular anomaly contains somatic MAP2K1 and KRAS mutations. Angiogenesis. 2019 Nov;22(4):547-552. doi: 10.1007/s10456-019-09678-w. Epub 2019 Sep 5. PMID 31486960
- [Background] Zeiser R, Andrlova H, Meiss F. Trametinib (GSK1120212). Recent Results Cancer Res. 2018;211:91-100. doi: 10.1007/978-3-319-91442-8_7. PMID 30069762
- [Background] Hashemzadeh S, Ramezani F, Rafii-Tabar H. Study of Molecular Mechanism of the Interaction Between MEK1/2 and Trametinib with Docking and Molecular Dynamic Simulation. Interdiscip Sci. 2019 Mar;11(1):115-124. doi: 10.1007/s12539-018-0305-4. Epub 2018 Nov 21. PMID 30465279
- [Background] Wright CJ, McCormack PL. Trametinib: first global approval. Drugs. 2013 Jul;73(11):1245-54. doi: 10.1007/s40265-013-0096-1. PMID 23846731
- [Background] Green JS, Norris DA, Wisell J. Novel cutaneous effects of combination chemotherapy with BRAF and MEK inhibitors: a report of two cases. Br J Dermatol. 2013 Jul;169(1):172-6. doi: 10.1111/bjd.12279. PMID 23413975
- [Background] Lekwuttikarn R, Lim YH, Admani S, Choate KA, Teng JMC. Genotype-Guided Medical Treatment of an Arteriovenous Malformation in a Child. JAMA Dermatol. 2019 Feb 1;155(2):256-257. doi: 10.1001/jamadermatol.2018.4653. PMID 30566190
- [Background] Adams DM, Trenor CC 3rd, Hammill AM, Vinks AA, Patel MN, Chaudry G, Wentzel MS, Mobberley-Schuman PS, Campbell LM, Brookbank C, Gupta A, Chute C, Eile J, McKenna J, Merrow AC, Fei L, Hornung L, Seid M, Dasgupta AR, Dickie BH, Elluru RG, Lucky AW, Weiss B, Azizkhan RG. Efficacy and Safety of Sirolimus in the Treatment of Complicated Vascular Anomalies. Pediatrics. 2016 Feb;137(2):e20153257. doi: 10.1542/peds.2015-3257. Epub 2016 Jan 18. PMID 26783326
- [Background] Steiner JE, Drolet BA. Classification of Vascular Anomalies: An Update. Semin Intervent Radiol. 2017 Sep;34(3):225-232. doi: 10.1055/s-0037-1604295. Epub 2017 Sep 11. PMID 28955111